CLINICAL TRIAL: NCT05892718
Title: A Phase 1, Open-label, Multi-center, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of HCB101 in Subjects With Advanced Solid Tumors or Relapsed and Refractory Non-Hodgkin Lymphoma
Brief Title: A Safety and Efficacy Study of HCB101, Fc-fusion Protein Targeting SIRPα-CD47 Pathway, in Solid or Hematological Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FBD Biologics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCB101-101
Record Dates: First submitted 2023-05-09; First posted 2023-06-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Refractory Non-Hodgkin Lymphoma
Keywords: Immunotherapy; CD47; SIRPα; Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HCB101 (Experimental): HCB101 in subjects with advanced solid tumors or relapsed and refractory non-Hodgkin lymphoma.
  Dosage levels: 0.08 mg/kg, 0.16 mg/kg, 0.32 mg/kg, 0.64 mg/kg, 1.28 mg/kg, 2.56 mg/kg, 5.12 mg/kg, 8.00 mg/kg, 12.00 mg/kg, 18.00 mg/kg, 24.00 mg/kg, 30.00 mg/kg and 36 mg/kg sequentially.
  Interventions: Drug: HCB101

INTERVENTIONS:
Drug: HCB101 — HCB101 administered via. intravenous (IV) infusion.
  Other Names: SIRPα-Fc fusion protein

SUMMARY:
The purpose of this study is to find out whether IV injection of HCB101 is an effective treatment for different types of advanced solid tumors or relapsed and refractory non-Hodgkin lymphoma and what side effects (unwanted effects) may occur in subjects aged 18 years old and above.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation, Phase 1 study. This study is to evaluate the safety, tolerability, pharmacokinetics (PK), anti-tumor activity, and identification of maximum tolerated dose (MTD) of HCB101 intravenous injection in adults with advanced solid tumors or relapsed and refractory non-Hodgkin lymphoma.

Eligible subjects must have failed standard therapies, been intolerable, or been considered medically inappropriate by the investigator. Subjects will be treated until unacceptable AEs, radiographic or clinical documented disease progression, withdrawal of consent, loss to follow-up, death, or termination of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Male and female subjects of ≥18 years of age.
3. Histologically/cytologically confirmed, locally advanced solid tumor: subjects with histologically or cytologically confirmed advanced solid tumors refractory to standard therapy, or for which no standard treatment exists or non-Hodgkin lymphoma, relapsed or refractory to at least 2 prior lines of therapy.
4. For subjects with advanced solid tumor - must have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at baseline.
5. For subjects with non-Hodgkin lymphoma - must have non-Hodgkin lymphoma that is measurable or assessable for response per Lugano Classification (with 2016 refinement).
6. Must have ECOG performance status of 0 to 2 at Screening.
7. Able to provide tumor tissue samples.
8. Have life expectancy of ≥12 weeks.

Exclusion Criteria:

1. With known history of hypersensitivity to any components of HCB101.
2. Known active or untreated CNS metastases and/or carcinomatous meningitis.
3. Have undergone a major surgery or radical radiotherapy or palliative radiotherapy or have used a radioactive drug that is not completed at least 2 weeks prior to the first dose of HCB101.
4. Clinically significant cardiovascular condition.
5. Any previous treatment-related toxicities which have not recovered to ≤ Grade 1 as evaluated by National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or baseline, except alopecia and anemia.
6. With known inherited or acquired bleeding disorder or bleeding diathesis. .
7. Have RBC transfusion within 4 weeks prior to Screening.
8. With a previously documented diagnosis of hemolytic anemia or Evans Syndrome in the last 3 months.
9. Any investigational or approved systemic cancer therapy.
10. Active use of vitamin K antagonist anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on case by case basis. There will be no restriction for daily aspirin ≤ 81 mg/QD.
11. Have used herbal medication within 14 days prior to the first dose of HCB101.
12. Have received any treatment targeting the CD47 or SIRPα pathway.
13. Have other malignancies requiring treatment within 2 years prior to the first dose of HCB101.
14. Participation in another clinical study with an investigational product administered in the last 14 days prior to receiving the first dose of HCB101.
15. An investigational device used within 28 days prior to the first dose of HCB101.
16. Positive for hepatitis B, active hepatitis C infections, positive for HIV, or known active or latent tuberculosis.
17. Known to have a history of alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Number/incidence and percentage of subjects with adverse events, including ADA. | 12 months
  To evaluate the safety and tolerability of HCB101
Number of subjects with MTD of HCB101 | 12 months
  To evaluate the safety and tolerability of HCB101

SECONDARY OUTCOMES:
Overall Rate Response (ORR) | 12 months
  ORR is defined as the proportion of participants who have a partial response (PR) or critical response (CR)
Duration of Response (DoR) | 12 months
  DOR is defined as time from date of initial documentation of a response (PR or CR) to date of first documented evidence of progressive disease (PD)
Disease Control Rate (DCR) | 12 months
  DCR is defined as the proportion of participants who have a partial response (PR), critical response (CR), or disease stable (SD)
Progression-Free Survival (PFS) | 12 months
  Defined as the duration from the start of treatment until tumor progression or death of any cause.
Peak Plasma Concentration (Cmax) of HCB101 | 12 months
  Peak Plasma Concentration (Cmax) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.
Area under the plasma concentration versus time curve (AUC) of HCB101 | 12 months
  Area under the plasma concentration versus time curve (AUC) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.
Time to maximum drug concentration in plasma (Tmax) of HCB101 | 12 months
  Time to maximum drug concentration in plasma (Tmax) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.
Terminal elimination half-life (t1/2) of HCB101 | 12 months
  Terminal elimination half-life (t1/2) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.

OTHER OUTCOMES:
CD47 receptor occupancy on circulating red blood cells (RBCs) | 12 months
  CD47 receptor occupancy on circulating red blood cells (RBCs) will be measured as an indication of target engagement.
Concentration of potential PD biomarkers in participants will be assess. | 12 months
  Changes in macrophage function related cytokines will be assess after HCB101 treatment.
ctDNA detection | 12 months
  ctDNA detection in participants using next-generation sequencing (NGS ).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Hematology-Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Carolina BioOncology, Huntersville, North Carolina
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China
- Taiwan (3):
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei